CLINICAL TRIAL: NCT00064103
Title: Clinical Protocol for Wild Type p53 Gene Induction in Premalignancies of Squamous Epithelium of the Oral Cavity and Oral Pharynx Via an Adenoviral Vector [NCI Supplied Agent Ad-p53, (INGN 201) (Advexin®) NSC 683550, IND# 7135]
Brief Title: Gene Therapy in Preventing Cancer in Patients With Premalignant Carcinoma of the Oral Cavity or Pharynx
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2012-02541; MDA-ID-00193; P50CA097007 (NIH); CDR0000306522 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Lip and Oral Cavity Cancer; Oropharyngeal Cancer; Stage 0 Lip and Oral Cavity Cancer; Stage 0 Oropharyngeal Cancer; Tongue Cancer
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Tongue Neoplasms | interventions — advexin

ARMS (1):
- Treatment (Ad5CMV-p53 gene) (Experimental): Phase I: Patients receive Ad5CMV-p53 gene by intramucosal injection into the area of the lesion followed at least 2 hours later by Ad5CMV-p53 gene as an oral rinse on day 1. Patients then receive Ad5CMV-p53 gene as an oral rinse twice daily on days 2-5. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of Ad5CMV-p53 gene as an oral rinse until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Phase II: Patients receive treatment with intramucosal Ad5CMV-p53 gene as in phase I and Ad5CMV-p53 gene as an oral rinse at the MTD.
  Interventions: Biological: Ad5CMV-p53 gene; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: Ad5CMV-p53 gene — Given intramucosally or as oral rinse
  Other Names: Ad5CMV-p53; ADVEXIN; INGN-201
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of gene therapy and to see how well it works in preventing cancer in patients with premalignant carcinoma of the oral cavity or pharynx. Inserting the p53 gene into a person's tumor cells may improve the body's ability to kill the tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the acute toxic effects of Ad5CMV-p53 gene administered as an oral rinse and as an intramucosal injection in patients with diffuse premalignant carcinoma of the oral cavity or oral pharynx.

II. Determine the maximum tolerated dose of this drug in these patients. III. Determine the topical transduction efficiency of adenoviral-mediated wild type p53 gene transfer in patients treated with this drug.

IV. Determine the efficacy of this drug in reversing the histology of oral premalignancies in these patients.

V. Determine the distribution of transgenic protein within the area of the premalignant lesion in patients treated with this drug.

OUTLINE: This is an open-label, dose-escalation study of Ad5CMV-p53 gene administered as an oral rinse.

Phase I: Patients receive Ad5CMV-p53 gene by intramucosal injection into the area of the lesion followed at least 2 hours later by Ad5CMV-p53 gene as an oral rinse on day 1. Patients then receive Ad5CMV-p53 gene as an oral rinse twice daily on days 2-5. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of Ad5CMV-p53 gene as an oral rinse until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Phase II: Patients receive treatment with intramucosal Ad5CMV-p53 gene as in phase I and Ad5CMV-p53 gene as an oral rinse at the MTD. Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years. Patients then receive long-term follow-up annually for an additional 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mild to moderate dysplasia OR severe dysplasia/carcinoma in situ of the oral cavity or oral pharynx

  * Clinically evident diffuse premalignant disease, defined by 1 of the following mucosal abnormalities:

    * Extension between adjacent organ structures (e.g., lateral tongue, ventral tongue, and the floor of the mouth)
    * Extensive surface area, including the entire ventral tongue or floor of the mouth or buccal mucosa, in a velvety "indiscreet" pattern
* Meets 1 of the following criteria:

  * Previously treated with conventional treatment (e.g., radiotherapy or surgery) for a prior head and neck malignancy
  * Failed biochemoprevention approaches for premalignant disease
  * Failed other therapeutic approaches for premalignant disease
* No active squamous cell carcinoma of the head and neck
* Performance status - Karnofsky 70-100%
* Absolute granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.0 mg/dL
* Creatinine no greater than 1.5 mg/dL
* No hypertension (baseline blood pressure 140/90 mm Hg or higher)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 1 year after study participation
* HIV-1 negative
* No known contact with former tissue or organ transplantation recipients or individuals with severe immunodeficiency disease (acquired or congenital) during and for 28 days after study treatment
* No prior malignancy within the past 2 years except nonmelanoma skin cancer or aerodigestive cancer
* No active systemic viral, bacterial, or fungal infections requiring treatment
* No serious concurrent illness that would preclude study compliance and follow-up
* No psychological, familial, sociological, geographical, or other condition that would preclude study compliance and follow-up
* See Disease Characteristics
* More than 21 days since prior chemotherapy (42 days for mitomycin and nitrosoureas)
* No concurrent systemic chemotherapy
* No concurrent prednisone or the equivalent, including corticosteroids of more than 10 mg/day
* See Disease Characteristics
* More than 3 months since prior radiotherapy involving the lesion selected for this study
* No concurrent radiotherapy
* See Disease Characteristics
* More than 8 weeks since prior investigational agents
* No prior experimental therapy (i.e., oral, systemic, topical, or direct injection) for the lesion selected for treatment in this study
* No other concurrent immunosuppressive therapy
* No other concurrent investigational agents
* No concurrent aspirin dose greater than 175 mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-06; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | Up to 15 years
Severity of adverse events graded using the CTCAE version 3.0 | Up to 15 years
Maximum tolerated dose of Ad5CMV-p53 gene | 6 months
  Evaluated by the frequency and relationship of dose-limiting toxicities, if any, experienced by patients during dose escalation.
Pharmacodynamics evaluated by examining the injected precancerous lesion for induction of apoptosis and expression of the p53 protein | 168 days
  Presented using descriptive statistics, frequency tabulations, and graphical displays over time by treatment cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Gary L. Clayman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States